CLINICAL TRIAL: NCT05693779
Title: Exercise Therapy After Pulmonary Thromboendarterectomy or Balloon Pulmonary Angioplasty for Chronic Thromboembolic Pulmonary Hypertension: EXPECT-PH
Brief Title: Exercise Therapy After Pulmonary Thromboendarterectomy or Balloon Pulmonary Angioplasty for Chronic Thromboembolic Pulmonary Hypertension
Acronym: EXPECT-PH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative Changes.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Brahmajee K Nallamothu, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00214495
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Exercise; Balloon pulmonary angioplasty; Pulmonary thromboendarterectomy; Smart watch; Treadmill exercise test
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home exercise training (Experimental): Individualized exercise prescription will be provided based on the gathered cardiopulmonary exercise test data.
  Interventions: Behavioral: Home exercise training

INTERVENTIONS:
Behavioral: Home exercise training — Participants will complete an Exercise Treadmill Test at baseline. The 12 weeks exercise program that will be assigned to each patient will be based on these results. The exercise will be three 20-minute exercise sessions per week for 6 weeks. This will increase to four 60-minute exercise sessions per week at increased intensity progressively over the course of the exercise program. The exercise program will involve walking/jogging, elliptical training, or biking 3-4 times per week for up to an hour each session. If participants don't have access to a bike or elliptical, they will be asked to exercise by walking/jogging.
  Participants will also a phone call or video chat that takes about 15 minutes per week to discuss the exercise program and take 2 short surveys weekly on the MyDataHelps application and filling out a logbook recording exercise sessions. In addition, participants activity will be measured by using a smartwatch during the study.

SUMMARY:
This study is being completed to determine the feasibility and acceptability of completing a home-based, structured, low-to-moderate intensity exercise training program in chronic thromboembolic pulmonary hypertension (CTEPH) patients following surgical or percutaneous intervention. Eligible participants will be enrolled and have a 12 week home based exercise training program.

The study team hypothesizes that:

The following percentage of participants successfully complete the ramp-up phase of the exercise program:

* Greater or equal to 70% at end of week 7
* Greater or equal to 80% at end of week 10
* Greater or equal to 90% at end of week 12
* Greater or equal to 80% of participants will both complete ≥1 week of maintenance phase exercise and complete 12 weeks of the exercise intervention.
* Patients will have no adverse events, defined as syncope, worsening World Health Organization (WHO) functional class, pulmonary hypertension (PH) related hospitalization, or death, caused by the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Thromboembolic Pulmonary Hypertension (CTEPH) patients post-Pulmonary Thromboendarterectomy (PTE) or Balloon Pulmonary Angioplasty (BPA)
* Planned follow-up at Michigan Medicine for at least one year
* Has access to an Android or iPhone with study supported operating software, is willing to install MyDataHelps application, and is willing to wear a smart watch while awake

Exclusion Criteria:

* Life expectancy under 1 year
* Orthopedic, neurological, or psychiatric condition limiting ability to actively engage in exercise training session
* Currently receiving palliative care and/or in hospice care
* Persistent severe Right Ventricular (RV) dysfunction on echocardiography post BPA or PTE
* Recently completed, current enrollment, or planned enrollment in pulmonary rehabilitation
* Moderate or severe obstructive lung disease or restrictive lung disease
* Arterial oxygen saturation (SpO2) <88% during 6 minute walk test(6MWT) on baseline home oxygen prescription
* Wrist too large to wear a smart watch comfortably.
* Participant noted to wear smart watch for less than 8 hours per day prior to intervention.
* Determined to be unsafe for participation in exercise therapy as assessed by the clinical team.
* Those with mobility issues that are unable to complete 6MWT.
* Participant has sex minute walk distance (6MWD) greater or equal to 90% predicted at visit 1.
* Pregnancy or lactation
* Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who complete the ramp-up phase of the exercise program at end of week 7 of the intervention | Week 7
  Based on intervention weeks 1-7. Compliance data will be documented by participants in virtual exercise logs and reviewed weekly with the study team.
Percentage of participants who complete the ramp-up phase of the exercise program at end of week 10 of the intervention | Week 10
  Based on intervention weeks 1-10. Compliance data will be documented by participants in virtual exercise logs and reviewed weekly with the study team.
Percentage of participants who complete the ramp-up phase of the exercise program at end of week 12 of the intervention | Week 12
  Based on intervention weeks 1-12. Compliance data will be documented by participants in virtual exercise logs and reviewed weekly with the study team.

SECONDARY OUTCOMES:
Number of adverse events | 12 weeks
  These will be defined as hospitalization due to CTEPH-specific decompensation, worsening World Health Organization (WHO) functional class, syncope, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Aggarwal, MD, Principal Investigator — University of Michigan; Bramajee Nallamothu, MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No